CLINICAL TRIAL: NCT03995888
Title: A Phase 1, Open-label Study to Assess Safety, Biodistribution, and Internal Radiation Dosimetry of rhPSMA-7.3 (18F) Injection in Healthy Volunteers, and to Assess Safety and Investigate the Imaging Characteristics in Subjects With Prostate Cancer
Brief Title: Assessing Radio-hybrid Prostate Specific Membrane Antigen (rhPSMA-7.3) (18F) in Healthy Volunteers and Subjects With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: BED-PSMA-101
Record Dates: First submitted 2019-06-18; First posted 2019-06-24 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Positron Emission Tomography (PET) Imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  Interventions: Drug: rhPSMA-7.3 (18F) Injection
- Patients (Experimental): Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  Interventions: Drug: rhPSMA-7.3 (18F) Injection

INTERVENTIONS:
Drug: rhPSMA-7.3 (18F) Injection — Radioligand for PET CT scanning

SUMMARY:
A Phase 1, Open-label Study to Assess Safety, Biodistribution, and Internal Radiation Dosimetry of rhPSMA-7.3 (18F) Injection in Healthy Volunteers, and to Assess Safety and Investigate the Imaging Characteristics in Subjects With Prostate Cancer.

ELIGIBILITY:
Key Inclusion Criteria: Healthy Volunteers

1. Male and females 21-65 years.
2. Clinically acceptable medical history

Key Exclusion Criteria: Healthy Volunteers

1. Received ionising radiation exposure from clinical trials or medical examinations or treatment in the last 12 months.
2. Suffers from claustrophobia.
3. Bilateral hip prostheses.

Key Inclusion Criteria: Patients

1. Male 18-80 years.
2. Histologically confirmed adenocarcinoma of the prostate
3. Clinically acceptable medical history
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Key Exclusion Criteria: Patients

1. Biopsy 28 days prior to enrollment.
2. Extensive metastatic disease.
3. Underlying disease which might confound interpretation.
4. Bilateral hip prostheses.
5. High energy (>300 Kiloelectron Volt (keV)) gamma-emitting radioisotope administered within five physical half-lives, or any intravenous iodinated contrast medium within 24 hours, or any high density oral contrast medium (oral water contrast is acceptable) within 5 days prior to study drug administration.
6. X-ray contrast agent (<24 hr for intravenous agents and <5 days for oral agents).
7. History of claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, Principal Investigator — Clinical Research Services Turku - CRST Oy
Locations (1):
- Clinical Research Services Turku - CRST Oy, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malaspina S, Oikonen V, Kuisma A, Ettala O, Mattila K, Bostrom PJ, Minn H, Kalliokoski K, Postema EJ, Miller MP, Scheinin M. Kinetic analysis and optimisation of 18F-rhPSMA-7.3 PET imaging of prostate cancer. Eur J Nucl Med Mol Imaging. 2021 Oct;48(11):3723-3731. doi: 10.1007/s00259-021-05346-8. Epub 2021 Apr 12. PMID 33846844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 11 June 2019 (first subject, screening visit) and 16 April 2020 (last subject, last visit) at a single site in Finland. Of the 24 potential subjects screened, 16 met all the study eligibility criteria (six healthy volunteers and 10 subjects with prostate cancer). Five subjects were considered screen failures and three subjects were not assigned to IMP as they were back-up subjects who were subsequently not required for PET imaging.
Pre-assignment Details: Baseline safety evaluations performed at screening (visit 1) comprised of vital signs, urine analysis, blood sample collection, pregnancy testing, physical exam, and recording of any adverse events (AEs) from the time of informed consent. Pertinent medical history and concomitant medications were also captured.
Groups:
- Prostate Cancer Cohort A: Subjects with unfavourable intermediate-risk or high-risk primary prostate cancer
  Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  rhPSMA-7.3 (18F) Injection: Radioligand for PET CT scanning
- Prostate Cancer Cohort B: Subjects with hormone-sensitive metastatic prostate cancer
  Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  rhPSMA-7.3 (18F) Injection: Radioligand for PET CT scanning
- Prostate Cancer Cohort C: Subjects with castration-resistant metastatic disease
  Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  rhPSMA-7.3 (18F) Injection: Radioligand for PET CT scanning
Period: Overall Study
Arm/Group | Healthy Volunteers | Prostate Cancer Cohort A | Prostate Cancer Cohort B | Prostate Cancer Cohort C
Started | 6 | 3 | 3 | 4
Completed | 6 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: Healthy Volunteers
  Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  rhPSMA-7.3 (18F) Injection: Radioligand for PET CT scanning
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Prostate Cancer Cohort A | Prostate Cancer Cohort B | Prostate Cancer Cohort C | Total
Number analyzed (Participants) | 6 | 3 | 3 | 4 | 16
Age, Continuous [Median (Full Range); unit: Years] | 62 [25 to 64] | 55 [55 to 56] | 69 [67 to 80] | 73 [65 to 76] | 64 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 4 | 13
  Male | 3 | 0 | 0 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 3 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Finland | 6 | 3 | 3 | 4 | 16
Height (cm [Median (Full Range); unit: Centimeters (cm)] | 175.25 [160 to 186] | 177.50 [172 to 180] | 174 [172 to 176.5] | 171.75 [160 to 184] | 173.27 [160 to 186]
Weight (kg) [Median (Full Range); unit: Kilograms (kg)] | 79.15 [66.5 to 89.8] | 81.80 [71.0 to 87.5] | 82.70 [75.5 to 83.5] | 79.40 [77.5 to 99.0] | 80.50 [66.5 to 99.0]
Body Mass Index (kg/m2) [Median (Full Range); unit: Kilograms/meters squared [kg^m2]] | 25.25 [23.2 to 30.0] | 27.70 [21.8 to 27.8] | 26.50 [25.5 to 27.6] | 28.45 [26.0 to 30.4] | 27.05 [21.8 to 30.4]
Eastern Cooperative Oncology Group (ECOG) [Number; unit: participants] — ECOG clinical gradings reported are described below. As grading number increases, participants are clinically considered as being less able to care for themselves, daily activity, and physical ability (walking, working, etc.).
  Grade 0: Fully active, able to carry on all pre-disease performance without restriction
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work Population: ECOG was not reported for those six participants in the 'Healthy Volunteers' cohort. Therefore, is entered as '0 participants analyzed'.
  participants
    0: number analyzed (Participants) | 0 | 3 | 3 | 4 | 10
    0 |  | 3 | 3 | 2 | 8
    1: number analyzed (Participants) | 0 | 3 | 3 | 4 | 10
    1 |  | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events as Classified by MedDRA
Description: Safety will be assessed from data on the occurrence of one or more treatment-emergent Adverse Events from the time of intravenous administration of 18F-rhPSMA-7.3 throughout the study period, and changes in serum biochemistry, hematology, coagulation, urinalysis, vital signs, Electrocardiogram (ECG), injection site status, and physical examination findings.
Time Frame: 1 month
Population: Participants who have received at least one dose of Flourine-18 radiohybrid prostate-specific membrane antigen-7,3.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers | Prostate Cancer Cohort A | Prostate Cancer Cohort B | Prostate Cancer Cohort C
Number analyzed (Participants) | 6 | 3 | 3 | 4
Participants | 2 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: As specified in the Statistical Analysis Plan, results are presented as only those treatment-emergent adverse events which occurred up to 1 Month after the 18F administration
Arm/Group | Healthy Volunteers | Prostate Cancer Cohort A | Prostate Cancer Cohort B | Prostate Cancer Cohort C
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/3 | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 2/6 | 1/3 | 1/3 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=6) | Prostate Cancer Cohort A (N=3) | Prostate Cancer Cohort B (N=3) | Prostate Cancer Cohort C (N=4)
Retention of urine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=6) | Prostate Cancer Cohort A (N=3) | Prostate Cancer Cohort B (N=3) | Prostate Cancer Cohort C (N=4)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT03995888/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03995888/SAP_001.pdf